CLINICAL TRIAL: NCT04838561
Title: Assessing the Impact of Control-IQ Technology on Quality of Life and Glycemic Control in Children and Youth With Type 1 Diabetes in a Canadian Context
Brief Title: Assessing the Impact of Control-IQ Technology
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Principal Investigator, Caroline Zuijdwijk, Pediatric Endrocinologist, MD FRCPC, Children's Hospital of Eastern Ontario
Other Study IDs: 21/26X
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-centre, mixed-methods, prospective study in pediatric patients with T1D initiating Control-IQ technology on the Tandem t-slim X2 insulin pump.

Primary Objective:

To determine pediatric T1D patients' and their parents' perceptions of the impact of Control-IQ on their psychosocial functioning and quality of life.

DETAILED DESCRIPTION:
Background Information & Rationale

The management of type 1 diabetes (T1D) is rapidly evolving to offer technology that aims to improve metabolic control and decrease the burden of diabetes management. Hybrid-closed loop systems are at the forefront of this technology. They are comprised of an insulin pump and continuous glucose monitoring (CGM) system that interface in order to automatically adjust the delivery of basal insulin through the pump, based on CGM data. Insulin boluses for meals and snacks must still be entered manually by the user.

Studies of hybrid closed loop systems have primarily focused on clinical trials that show improved glycemic outcomes.1-3 Few studies have assessed real-world glycemic outcomes or patient-reported outcomes, and none have focused on a pediatric population.

A recent study published by Pinsker et al.4 showed improvement in psychosocial outcomes and persistent achievement of glycemic targets in a real-world setting in adults with T1D using the Tandem t:slim X2 pump with Control-IQ technology.

The Tandem t:slim X2 pump with Control-IQ is a hybrid closed loop system (using Dexcom G6 CGM) that has recently been approved for use by Health Canada, but has been used in the U.S. for the last year. This new technology will launch in Canada in March 2021, at which time existing Tandem t:slim X2 insulin pump users (with concurrent CGM use) will be able to upgrade their insulin pump software to access this technology (following review of an online module).

The Children's Hospital of Eastern Ontario (CHEO), is located in Ottawa, ON Canada. CHEO follows approximately 800 children with diabetes, approximately 85 of whom are managed on the Tandem t:slim X2 pump with concurrent Dexcom G6 CGM use.

The upcoming launch of Control-IQ presents a unique opportunity to gain a better understanding of the real-world impact of this technology on our Canadian pediatric population. The benefits of conducting this study in our population are two-fold:

1. The Canadian context offers the study a diverse patient population given our universal healthcare system and provincially-funded insulin pump program. Because pumps and supplies are funded by the government, they are available to all of our patients, regardless of socio-economic status and whether or not they have private health insurance.
2. Studying a pediatric population offers the unique perspective of children and youth (and their parents) whose management practices and goals differ from those of adults. While adult patients and parents of children with T1D are motivated by attaining glycemic targets for long term health outcomes, children and youth live in moment with emphasis on how they feel now. As such, patient reported outcomes, while important to all ages, are often the most important motivator for children and youth when choosing a treatment regimen.

Study Design This is a single-centre, mixed-methods, prospective study in pediatric patients with T1D initiating Control-IQ technology on the Tandem t-slim X2 insulin pump.

Participants will enroll in the study prior to initiating use of Control-IQ on their Tandem insulin pump.

Recruitment will occur over an eight-week period starting mid-March 2021. Participation in this study will last 16 weeks.

Study Objectives

Primary Objective: To determine pediatric T1D patients' and their parents' perceptions of the impact of Control-IQ on their psychosocial functioning and quality of life (as measured by the INSPIRE Questionnaire, post assessment).

Secondary Objectives:

1. To assess the effect of Control-IQ technology on other patient and parent reported outcomes (PROs) including:

   * Diabetes Impact and Device Satisfaction (DIDS) scale,
   * Hypoglycemia Fear Survey (child and parent version),
   * WHO-5 (emotional well-being)
2. To determine the impact of Control-IQ technology on glycemic control in pediatric T1D patients who are experienced sensor-augmented pump users.

Exploratory Objectives:

1. To explore the effect of Control-IQ technology on patient and parents' sleep, school, activities/ sports, mood and family dynamics.
2. To explore whether or not youth and parents' expectations of Control-IQ align with their experience of using this this automated insulin delivery system.

Participant Characteristics:

The following data will be collected from each chart at baseline:

* Date of birth
* Gender
* Date of T1D diagnosis
* Date of initiation of insulin pump therapy

  * Date of first insulin pump start
  * Date of Tandem t:slim X2 pump start
* Current use of CGM (yes/ no)
* Last measured HbA1c ( if available within the last 3 months
* Number of hospitalizations due to diabetes complications within the past year

Sociodemographic measures will be collected by questionnaire at baseline, including:

* Family structure
* Parental education - highest level achieved
* Household income
* Private health insurance
* Ethnicity (self-reported)

Statistical Plan The patient population will be described using descriptive statistics. The study team will compare patient reported outcomes, measures of glycemic control, and measures of insulin pump management pre and 16 weeks post-initiation of Control-IQ technology, using paired t-test and Wilcoxon signed-rank test, depending on the distributional characteristics of the outcomes. Analysis of open-ended questions will be done by a qualitative research specialist.

Sample Size Determination CHEO currently has 85 patients on the Tandem t:slim X2 pump with CGM, with an estimated 10-15 patients more estimated to start before March 2021. Historically, the patient population at CHEO has been highly engaged with research with an anticipated participation rate of 90-95%. The Investigator expects that recruitment rates would be similar for this study, allowing for a sample size of 70 participants.

This sample size is sufficient to provide > 80% power for detecting a "medium size" effect (Cohen's d = 0.5), which corresponds to a mean score of 70 from the post assessment INSPIRE Questionnaire, 10 units larger than a mean score of 60 (the null hypothesis). Cohen's d is expressed by the ratio of the mean difference over the standard deviation. Here, we use sd = 20 as an estimate of the standard deviation of the score, which is conservative considering previously presented estimates (e.g. sd = 16.44 described in Weissberg-Benchell et al [5]).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of T1D
2. Age 6-18 years
3. Currently using the Tandem t:slim X2 insulin pump with Dexcom G6 CGM, who are initiating Control-IQ

Exclusion Criteria:

1. Patients under the age of 6 years of age
2. Patients who are not English or French speaking
3. Patients unwilling to provide consent (assent where applicable).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and youth with T1D followed at CHEO will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
INsulin delivery Systems: Perceptions, Ideas, Reflections and Expectations Questionnaire Post Intervention (Youth and Parent Versions) | 16 weeks
  Measures perceptions of the impact of automated insulin delivery systems on users' psychosocial functioning and quality of life.
  Score 0-100- mean score is significantly larger than 60 (out of 100). A score of greater than 60 indicates a perceived benefit of Control-IQ on psychosocial functioning and quality of life.

SECONDARY OUTCOMES:
Change in Diabetes Impact and Device Satisfaction scale | Baseline and 16 weeks
  Evaluates users' experience interacting with their insulin delivery device, and the impact of diabetes on their life on a 10-point Likert Scale. Scoring: Device Satisfaction average of items 1-7 (#5, #7 are reverse scored), Diabetes Impact: Average of items 8-11. Higher Score Indicates increased device satisfaction.
Hypoglycemia Fear Survey (child and parent version) | Baseline and 16 weeks
  Assess change in fear of hypoglycemia among children with type 1 diabetes and parents of children with type 1 diabetes.
  Mean score will be compared pre and post study Behaviour (score 0-40) - lower score better (less behaviours associated with fear of hypo) Worry (score 0-60) - lower score better (less worry re: hypoglycemia)
The World Health Organisation- Five Well-Being Index | Baseline and 16 weeks
  Assessing change in subjective psychological well-being in research and clinical settings.
  The WHO-5 consists of five statements, which respondents rate according to the scale below (in relation to the past two weeks).
  * All of the time = 5
  * Most of the time = 4
  * More than half of the time = 3
  * Less than half of the time = 2
  * Some of the time = 1
  * At no time = 0.
  The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
% time in target range 3.9-10.0 mmol/L (overall, day,and night) | 0, 4, 8, 12, and 16 weeks
  Measure of glycemic control will be collected from the Dexcom Clarity Platform will be compared at each time frame.
% time below target range <3.0mmol/L (overall, day, and night) | 0, 4, 8, 12, and 16 weeks
  Measure of glycemic control will be collected from the Dexcom Clarity Platform will be compared at each time frame.
% time below target range <3.9mmol/L (overall, day, and night) | 0, 4, 8, 12, and 16 weeks
  Measure of glycemic control will be collected from the Dexcom Clarity Platform will be compared at each time frame.
% time above target range >10mmol/L (overall, day, and night) | 0, 4, 8, 12, and 16 weeks
  Measure of glycemic control will be collected from the Dexcom Clarity Platform will be compared at each time frame..
% time above target range >13.9mmol/L (overall, day, and night) | 0, 4, 8, 12, and 16 weeks
  Measure of glycemic control will be collected from the Dexcom Clarity Platform will be compared at each time frame.
Average glucose and standard deviation (mmol/L) | 0, 4, 8, 12, and 16 weeks
  Measure of glycemic control will be collected from the Dexcom Clarity Platform will be compared at each time frame.
Coefficient of variation (%) | 0, 4, 8, 12, and 16 weeks
  Measure of glycemic control will be collected from the Dexcom Clarity Platform.
Estimated HbA1c (%) | 0, 4, 8, 12, and 16 weeks
  Will be collected from the Dexcom Clarity Platform.

OTHER OUTCOMES:
Open-Ended Questionnaire | 16 weeks
  Explores the effect of Control-IQ technology on patient and parents' sleep, school, activities/ sports, mood and family dynamics
INsulin delivery Systems: Perceptions, Ideas, Reflections and Expectations Questionnaire (Baseline and Post Intervention) | Baseline and 16 weeks
  To explore whether or not youth and parents' expectations of Control-IQ align with their experience of using this this automated insulin delivery system (by comparing the INSPIRE Questionnaire baseline and post-assessment scores)
  Score 0-100- mean score is significantly larger than 60 (out of 100). A score of greater than 60 indicates a perceived benefit of Control-IQ on psychosocial functioning and quality of life.
  Mean baseline INPSIRE score will be compared to the mean post-assessment INSPIRE score to assess if expectations of Control-IQ align with the experience of using this automated insulin delivery system.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Zuijdwijk, MD, FRCPC, Principal Investigator — Children's Hopsital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Malley G, Messer LH, Levy CJ, Pinsker JE, Forlenza GP, Isganaitis E, Kudva YC, Ekhlaspour L, Raghinaru D, Lum J, Brown SA; iDCL Trial Research Group. Clinical Management and Pump Parameter Adjustment of the Control-IQ Closed-Loop Control System: Results from a 6-Month, Multicenter, Randomized Clinical Trial. Diabetes Technol Ther. 2021 Apr;23(4):245-252. doi: 10.1089/dia.2020.0472. PMID 33155824
- [Background] Brown SA, Kovatchev BP, Raghinaru D, Lum JW, Buckingham BA, Kudva YC, Laffel LM, Levy CJ, Pinsker JE, Wadwa RP, Dassau E, Doyle FJ 3rd, Anderson SM, Church MM, Dadlani V, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Kollman C, Beck RW; iDCL Trial Research Group. Six-Month Randomized, Multicenter Trial of Closed-Loop Control in Type 1 Diabetes. N Engl J Med. 2019 Oct 31;381(18):1707-1717. doi: 10.1056/NEJMoa1907863. Epub 2019 Oct 16. PMID 31618560
- [Background] Dadlani V, Pinsker JE, Dassau E, Kudva YC. Advances in Closed-Loop Insulin Delivery Systems in Patients with Type 1 Diabetes. Curr Diab Rep. 2018 Aug 29;18(10):88. doi: 10.1007/s11892-018-1051-z. PMID 30159816
- [Background] Pinsker JE, Muller L, Constantin A, Leas S, Manning M, McElwee Malloy M, Singh H, Habif S. Real-World Patient-Reported Outcomes and Glycemic Results with Initiation of Control-IQ Technology. Diabetes Technol Ther. 2021 Feb;23(2):120-127. doi: 10.1089/dia.2020.0388. Epub 2020 Sep 10. PMID 32846114
- [Background] Weissberg-Benchell J, Shapiro JB, Hood K, Laffel LM, Naranjo D, Miller K, Barnard K. Assessing patient-reported outcomes for automated insulin delivery systems: the psychometric properties of the INSPIRE measures. Diabet Med. 2019 May;36(5):644-652. doi: 10.1111/dme.13930. Epub 2019 Mar 20. PMID 30761592
- [Background] Cox DJ, Irvine A, Gonder-Frederick L, Nowacek G, Butterfield J. Fear of hypoglycemia: quantification, validation, and utilization. Diabetes Care. 1987 Sep-Oct;10(5):617-21. doi: 10.2337/diacare.10.5.617. PMID 3677982
- [Derived] Zuijdwijk C, Courtney J, Mitsakakis N, Hayawi L, Sutherland S, Newhook D, Ahmet A, Goldbloom EB, Khatchadourian K, Lawrence S. Control-IQ Technology Positively Impacts Patient Reported Outcome Measures and Glycemic Control in Youth with Type 1 Diabetes in a Real-World Setting. Pediatr Diabetes. 2023 Apr 12;2023:5106107. doi: 10.1155/2023/5106107. eCollection 2023. PMID 40303267